CLINICAL TRIAL: NCT03009552
Title: Speckle Tracking Echocardiography Adds Information in Decompensated Heart Failure
Acronym: STRAIN-DHF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marco Stephan Lofrano Alves (Other)
Responsible Party: Sponsor-Investigator, Marco Stephan Lofrano Alves, MD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: CAAE:59669416.0.0000.0068; 2015/10005-5 (Other Grant/Funding Number: Sao Paulo Research Foundation)
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Decompensated Heart Failure
Keywords: speckle tracking echocardiography; strain; strain rate; torsion
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: speckle tracking echocardiography — Speckle tracking echocardiography is used for measuring parameters of cardiac mechanics: left ventricle strain and strain rate; left ventricle twist, untwist and torsion; left atrium strain and strain rate; right ventricle longitudinal strain and strain rate. Echocardiography will be performed within 24 hours of admission, 72 hours after admission and 1 month after discharge.

SUMMARY:
The overall objective of the study is to determine whether speckle tracking echocardiography presents additional prognostic value to the routine assessment (clinical and echocardiographic) in patients admitted with acute decompensated heart failure (ADHF) at the emergency department. Specific objectives: 1 - To evaluate the association between changes in the cardiac contractile mechanics (by serial measurements of strain, strain rate, displacement velocity, rotation and ventricular torsion) with clinical outcomes in ADHF. 2 - Evaluate the possible association of these parameters with biomarkers of neurohormonal activity, myocardial injury, fibrosis and myocardial remodeling, inflammatory activity, and cardiorenal syndrome.

DETAILED DESCRIPTION:
ADHF syndromes comprise around one million of emergency admissions per year in the United States, and the number of cases tripled in the last three decades, currently representing the main cause of hospital admission in patients over the age of 65 years. A recent study showed that among patients with similar risk in the presentation of ADHF, those admitted and treated in the emergency (in attempt to get early discharge) have higher mortality rate than those treated by hospitalization. On the other hand, uncertainty about the clinical course can also result in prolonged and unnecessary hospitalizations, which burdens the health system and consumes resources. Thus, It is vital to carry out studies that bring a better understanding of the pathophysiology of ADHF and to determine new risk stratification tools in the emergency department. Echocardiography is the most widely used imaging method and has a key role in the diagnosis and management of patients with HF. However, some methodological limitations of conventional echocardiography cause low reproducibility and intra and inter-observer agreement for some parameters, reducing their prognostic ability. In recent years, new technologies have been incorporated into the method in an attempt to overcome these limitations. One of these new technologies is echocardiography with "speckle tracking". The method, by its nature, has a significant advantage over parameters derived from conventional echocardiography, because of its ultrasound beam angle-independence. However, there is a paucity of data on this new technology in patients with ADHF in literature and we have not found studies evaluating the prognostic value of this method in a prospective cohort of patients in this condition. This study aims to develop knowledge of this assessment tool for cardiac mechanics in emergency care, exploring its potential prognostic value in patients with ADHF, aiming to assist the cardiologist in identifying eligible patients for early and safe discharge, and to identify those patients for whom hospitalization and longer treatment are recommended.

ELIGIBILITY:
Inclusion Criteria:

* Admission in the emergency for decompensated heart failure.

Exclusion Criteria:

* Systolic blood pressure < 85, need surgical treatment, high ventricular frequency atrial fibrillation or flutter, severe pulmonary disease, pulmonary embolism, septic shock, advanced malignant neoplasia, pregnancy, heart transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Decompensated heart failure
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of mortality, heart transplant, left ventricular assist device and readmission for decompensated heart failure. | Six months after admission

SECONDARY OUTCOMES:
Development of cardio-renal syndrome (loss of more than 30% of calculated creatinine clearance or need for dialysis) | 1 month after admission
Cardiac mortality | 6 months

OTHER OUTCOMES:
Changes in left ventricle strain | 72 hours after admission
Changes in left ventricle strain rate | 72 hours after admission
Changes in left ventricle torsion | 72 hours after admission
Changes in left ventricle ejection fraction | 72 hours after admission
Changes in left atrial strain | 72 hours after admission
Changes in left atrial strain rate | 72 hours after admission
Changes in left atrial volume | 72 hours after admission
Changes in right ventricle longitudinal strain | 72 hours after admission
Changes in right ventricle longitudinal strain rate | 72 hours after admission
Changes in right ventricle fractional area change | 72 hours after admission
Changes in right ventricle performance index | 72 hours after admission
Changes in right ventricle contraction-pressure index | 72 hours after admission
Changes in right ventricle load adaptation index | 72 hours after admission
Changes in tricuspid annular plane systolic excursion | 72 hours after admission
Changes in tricuspid tissue Doppler peak systolic velocity (s´) | 72 hours after admission
Changes in biventricular strain index | 72 hours after admission
Serum level of B-type natriuretic peptide (BNP) | 72 hours after admission
Serum levels of troponin | 72 hours after admission
Serum levels of Neutrophil gelatinase-associated lipocalin (NGAL) | 72 hours after admission
Serum levels of galectin-3 | 72 hours after admission
Serum levels of C-reactive protein | 72 hours after admission

CONTACTS AND LOCATIONS:
Overall Officials: Marco Stephan L Alves, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- CEPEC - Centro de pesquisas em ecocardiografia e cardiologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No